CLINICAL TRIAL: NCT04077710
Title: Safety and Efficacy of Three-dimensional Printing Template-assisted CT-guided Radioactive Iodine-125 Seeds Implantation in the Treatment of Recurrent Chest Wall Malignancies After External Beam Radiotherapy
Brief Title: RISI in the Treatment of Recurrent Chest Wall Malignancies After EBRT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CNRBG-2019-CWM-RISI
Record Dates: First submitted 2019-09-01; First posted 2019-09-04 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-05

CONDITIONS: Chest Wall Tumor
Keywords: radioactive iodine-125 seeds implantation; 3D-printing template; chest wall malignancies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Radioactive Iodine-125 Seeds Implantation — The radioactive Iodine-125 seed can release low dose of irradiation persistently which kills tumors cell and causes less damage to normal tissue at the same time. The treatment was performed under CT monitoring. 3D-printing template includes information on the path of the implantation needle, characteristics of the surface of the therapy area of the patient, and positioning and orientation effects which can make the operation more accurate.

SUMMARY:
This study will observe the efficacy and toxicities of 3-dimensional printing noncoplanar template assisted CT guided radioactive iodine-125 seeds implantation in the treatment of patients with recurrent chest wall malignancies after external beam radiotherapy prospectively, and analyzes the influence of clinical and dosimetric factors on the outcomes.

DETAILED DESCRIPTION:
Radioactive Iodine-125 seed brachytherapy is a conventional treatment in Peking University Third Hospital. Radioactive Iodine-125 seed brachytherapy is the implantation of Iodine-125 seed into tumors.The radioactive Iodine-125 seed can release low dose of irradiation persistently which kills tumors cell and causes less damage to normal tissue at the same time. This study will enroll the patients with recurrent chest wall malignancies after external beam radiotherapy (primary or metastasis) who underwent CT-guided radioactive iodine-125 seed implantation assisted by 3D-printing template from 2019 to 2021. The investigators evaluate the dose that covers 90% target volume(D90) and other parameters after the implantation. The efficacy and adverse events will be observed. Local control(LC) time and overall survival(OS) time are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* histological proven malignant tumor
* tumor located in chest wall and lesion diameter <= 10 cm
* recurrence after external beam radiotherapy
* there is no bleeding tendency
* there are no serious or uncontrolled underlying diseases (such as severe or uncontrolled hypertension, diabetes, cardiovascular and cerebrovascular diseases, and/or organ dysfunction
* there is an appropriate puncture path which is expected to achieve the treatment dose
* KPS > 70, which is expected to be able to tolerate puncture/ brachytherapy, and the expected survival time is longer than 3 months

Exclusion Criteria:

* there are skin ulceration, or with high risk of skin infection and ulceration
* liquefaction and necrosis in a large area in tumor with poor expected seeds distribution
* pregnant women, lactating women, psychiatric patients
* patients with poor compliance can not complete the treatment
* patients that researchers considered inappropriate to participate in this clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with chest wall malignancies (primary or metastasis) who were treated with CT-guided radioactive iodine-125 seeds implantation assisted by 3D-printing template during 2019 to 2021 will included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Local control time | Outcomes will be followed up every 2-3 months after enrollment. The total follow-up time is 3 years.
  The time from the date of seeds implantation to the date of recurrence of the implanted tumor or the date of last observation.
Incidence of adverse events | Outcomes will be followed up every 2-3 months after enrollment. The total follow-up time is 3 years.
  The adverse events are evaluated by the common terminology criteria for adverse events (CTCAE). The rate of each adverse event will be measured.

SECONDARY OUTCOMES:
Overall survival time | Outcomes will be followed up every 2-3 months after enrollment. The total follow-up time is 3 years.
  The time from the date of seeds implantation to the date of death from any cause or the date of last observation.

CONTACTS AND LOCATIONS:
Overall Officials: Junjie Wang, M.D. Ph.D, Principal Investigator — Department of Radiation Oncology, Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: CSR
Time Frame: Data will be available within 6 months of the study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.